CLINICAL TRIAL: NCT04491630
Title: COping With PAin Through Hypnosis, Mindfulness and Spirituality
Acronym: COPAHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida (Other)
Responsible Party: Principal Investigator, Maria Alexandra Ferreira Valente, Researcher, ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ISPA
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Pain, Acute
Keywords: Experimental pain; Self-hypnosis; Mindfulness meditation; Christian prayer
MeSH Terms: conditions — Acute Pain | interventions — Hypnosis; Mindfulness

STUDY DESIGN:
Intervention Model Description: A randomized 4-group, 196-subject experimental mixed-model repeated-measures study to:
  1. compare the immediate effects of self-hypnosis (SH), mindfulness meditation (MM), and Christian meditation (CM), relative to a control group (CN), for increasing pain tolerance and reducing pain intensity and pain-related stress, in response to experimental painful stimulation in a sample of healthy volunteers;
  2. to identify possible shared and unique predictors of response to the three treatment conditions.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and the experimenter who will conduct assessments and administer the audio-recorded interventions will be blind to the condition to which subjects will be assigned and to the study hypotheses. During informed consent, prospective participants will be told that they will listen to an audio-recording that previous research found to be helpful to pain management, and that the purpose of the study is to assess this the effects of this audio-recording on discomfort associated with the sensation of coldness. Participants will also be instructed not to disclose details of the content of the audios they receive to the experimenter. The research staff member responsible for participants' randomization will be blind to identifying information and to the code identifying each condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-Hypnosis (SH) (Active Comparator)
  Interventions: Behavioral: Self-Hypnosis (SH)
- Mindfulness meditation (MM) (Active Comparator)
  Interventions: Behavioral: Mindfulness Meditation (MM)
- Christian prayer (CP) (Active Comparator)
  Interventions: Behavioral: Christian Prayer (CP)
- Control condition (CN) (No Intervention): Participants in the CN condition will not be instructed to use any particular coping strategy to cope with the painful stimulation provided by the Cold Pressor Arm Wrap. Participants in the CN condition will listen to a 20-minute natural history audio recording. The option for this recording is supported by: (a) previous research showing that individuals who were asked to listen to it found it to be a neutral, yet relaxing, passage; (b) the use of this passage as an effective control condition in previous studies.

INTERVENTIONS:
Behavioral: Self-Hypnosis (SH) — Participants assigned to this condition will listen to a 20-minute recording with instructions of SH adapted from one of our team member's proposed model. First, the audio recording will introduce and orient the participant to SH. Then instruction in SH will be provided, including: (a) how to self-induce a hypnotic induction; (b) specific self-suggestions for comfort and ability to manage intense sensations; and (c) post-hypnotic suggestions that the participant will be easily able to use these hypnotic strategies on their own at a later time (i.e., in this case, during the Cold Pressor Arm Wrap procedures that will follow).
  A second 5-minute audio recording with instructions to guide the participant in SH will be provided during the second cycle of Cold Pressor Arm Wrap (CPAW).
  Arms: Self-Hypnosis (SH)
Behavioral: Mindfulness Meditation (MM) — Participants in the MM condition will listen to a 20-minutes recording with instructions in the use and application of Vipassana MM, adapted from the manual developed by one of our team members. First, the audio recording will focus on introducing the idea of attention to their breath, and of non-judgmental monitoring and acceptance of the all events and stimuli. Then a guided MM (body scan) experience will be provided.
  A second 5-minute audio recording with instructions to facilitate the MM (body scan) experience taught in the first audio recording will be provided during the second cycle of CPAW.
  Arms: Mindfulness meditation (MM)
Behavioral: Christian Prayer (CP) — Participants in this condition will listen to a 20-minute recording with CP instructions. These instructions will be adapted from the existing on-line biblical meditations from the Society of Jesus (www.passo-a-rezar.net). First, the recording will introduce and orient the participant to CP. Then, a text of the Bible will be read twice, followed by a brief suggestion of prayer.
  A second 5-minute audio recording with instructions to facilitate the CP experience taught in the first audio recording, including the recording of a text of the Bible followed by a brief suggestion of meditation and relaxing music, will be provided during the second cycle of CPAW.
  Arms: Christian prayer (CP)

SUMMARY:
The purpose of this study is to evaluate and compare the immediate effects of self-hypnosis, mindfulness meditation and a spiritual intervention relative to a control condition for increasing pain tolerance and reducing pain intensity and pain-related stress, in response to experimental painful stimulation.

DETAILED DESCRIPTION:
The primary aim of this study (Aim 1) is to compare the immediate effects of self-hypnosis (SH), mindfulness meditation (MM), and Christian meditation (CM), relative to a control group (CN), for increasing pain tolerance and reducing pain intensity and pain-related stress, in response to experimental painful stimulation in a sample of healthy volunteers.

An exploratory aim of this study (Aim 2) is to identify possible shared and unique predictors of response to the three treatment conditions. The possible predictors we plan to test include sex, age, religious affiliation, hypnotic suggestibility, baseline mindfulness, acceptance, pain-related beliefs, religiosity, trait spirituality, previous experience with SH, MM and CP, outcome expectancies, and trait absorption.

This is a randomized quantitative experimental mixed-model repeated-measures study with three assessment points: baseline (T0), pre-test (T1), and post-test (T2). Eligible healthy adults will be randomized to one of the four study conditions. Interventions will be a 20-minutes audio-guided practice of either self-hypnosis, mindfulness meditation, or Christian prayer. Participants in the control group will not be instructed to use any specific strategy during the painful stimulation. Participants will be submitted to a first cycle of Cold Pressor Arm Wrap. They will then listen to a 20-minutes audio recording inducing one of the three interventions, or, in the case of the control group, to a 20-minutes recording of a natural history textbook. Primary outcomes are pain intensity, pain tolerance, and pain-related stress as measured by salivary cortisol level and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older;
* able to read, speak and understand Portuguese;
* willing to be randomly assigned to all four conditions (regardless of participant's own religious affiliation)

Exclusion Criteria:

* reporting history of musculoskeletal problems, cancer, heart disease, stroke, epilepsy, diabetes, or Raynaud syndrome;
* having an open wound, cut, or fracture in any of the upper limbs;
* self-reported alcohol or substance dependence;
* cognitive or physical impairment, or severe psychopathology that could prevent participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Pre-treatment (collected up to 30 minutes before intervention), and post-treatment (collected up to 30 minutes after intervention)
  0-10 Numerical Rating Scale
Change in Pain Tolerance | Pre-treatment (collected up to 30 minutes before intervention), and post-treatment (collected up to 30 minutes after intervention)
  Length (in seconds) that an individual bears painful stimulation

SECONDARY OUTCOMES:
Change in Pain-related stress (Heart rate) | Pre-treatment (collected up to 30 minutes before intervention), and post-treatment (collected up to 30 minutes after intervention)
  Heart rate
Change in Pain-related stress (Salivary cortisol level) | Pre-treatment (collected up to 30 minutes before intervention), and post-treatment (collected up to 30 minutes after intervention)
  Salivary cortisol level

OTHER OUTCOMES:
Hypnotic suggestibility | Baseline
  Barber Suggestibility Scale (BSS). Objective scoring ranges from 0 to 8, and the subjective score ranges from 0 to 24. Higher scores indicate higher levels of hypnotic suggestibility.
Baseline mindfulness | Baseline
  Five-Facet Mindfulness Questionnaire. This is a self-report questionnaire composed of 39 items divided in five domains (observing, describing, acting with awareness, non-judging, and non-reactivity). The items are answered in a 5-point Likert scale, from 0 ("never") to 4 ("always"). Higher scores indicate greater mindfulness capacities.
Acceptance | Baseline
  Acceptance and Action Questionnaire-II. The items of the 7-item AAQ-II are answered in a 7-point type of Likert scale (from 1 = "never true") to 7 ("always true") that assess a single domain of acceptance. Higher scores indicate higher degree of acceptance.
Pain-related beliefs | Baseline
  35-item Survey of Pain Attitudes (35-item SOPA). This is a 35-item self-report questionnaire assessing seven pain-related beliefs or domains: pain control, disability, medical cure, solicitude, medication, emotion, and harm. Participants are asked to specify their degree of agreement with each statement in a Likert scale from 0 ("This is very untrue for me") to 4 ("This is very true for me"). Seven scores (one per pain-related belief) are computed. Higher scores indicate greater agreement with each belief.
Trait spirituality | Baseline
  Spiritual Transcendence Scale. This is a 24-item self-report questionnaire assessing three domains: prayer fulfillment, universality and connectedness. Respondents are asked to rate their degree of agreement with each statement in a Likert scale, from 1 ("completely disagree") to 5 ("completely agree"). Higher scores indicate greater trait spirituality.
Religiosity | Baseline
  Duke University Religiosity Index. This is a 5 items measure that assesses three major dimensions (corresponding the scale's three domains or subscales) of religious involvement: organizational religious activity, non-organizational religious activity, and intrinsic or subjective religiosity. Two items are answered in a 6 points type of Likert scale, from 1 to 6. Three items are answered in a 5 points Likert scale, from 1 to 5. Higher scores on the three subscales and on the total score of the measure indicate higher religiosity.

CONTACTS AND LOCATIONS:
Locations (1):
- ISPA, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira-Valente A, Van Dyke BP, Day MA, Teotonio do Carmo C, Pais-Ribeiro J, Pimenta F, Costa RM, Jensen MP. Immediate Effects of Hypnosis, Mindfulness Meditation, and Prayer on Cold Pressor Outcomes: A Four-Arm Parallel Experimental Study. J Pain Res. 2022 Dec 23;15:4077-4096. doi: 10.2147/JPR.S388082. eCollection 2022. PMID 36582659
- [Derived] Ferreira-Valente A, Pimenta F, Costa RM, Day MA, Pais-Ribeiro J, Jensen MP. COPAHS Study: protocol of a randomised experimental study comparing the effects of hypnosis, mindfulness meditation, and spiritual practices on experimental pain in healthy adults. BMJ Open. 2021 Feb 8;11(2):e040068. doi: 10.1136/bmjopen-2020-040068. PMID 33558346